CLINICAL TRIAL: NCT06280911
Title: The Effect of Consumption of Date Fruit and Nipple Stimulation in Late Pregnancy on The First Stage of Labor
Brief Title: The Effect of Consumption of Date Fruit and Nipple Stimulation in Late Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Halime Esra Meram, Principal Investigator, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 098
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Augmentation; Induction; Labor; Stimulation, Self
Keywords: Augmentation; Date fruit; Induction; Labor; Nipple Stimulation
MeSH Terms: conditions — Self Stimulation

STUDY DESIGN:
Intervention Model Description: The study was designed to be randomly controlled.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Date fruit group (Experimental): * Pregnant women were asked to consume 6 (about 65 gr) per day of dry date (Medjoul species) provided by the researcher until the birth of the 37th gestational age.
  * Dry date fruit provided by the researcher was given to the women to consume (42 pieces per week).
  * It has been stated that pregnancies should end the consumption of dates when actual uterine contractions begin.
  * Within the first 24 hours of labor, information on labor was recorded in the delivery file and "structured information form".
  Interventions: Other: Date Fruit group
- Nipple group (Experimental): * The pregnancies are requested to stimulate a nipple (three minutes a day, one minute in the morning, one noon, one minute in the evening) and three minutes in the other nipple (one minute morning, one noon, one minute evening) with naked fingures and moderate pressure by pulling and rounding.
  * The pregnancies were stated to terminate the nipple stimulation when the actual uterine contractions onset.
  * Within the first 24 hours of labor, information on labor was recorded in the labor file and "structured information form".
  Interventions: Other: Nipple group
- Control group (No Intervention): • Within the first 24 hours of labor, information on labor was recorded in the delivery file and "structured information form".

INTERVENTIONS:
Other: Date Fruit group — Consumption of Date Fruit
  Arms: Date fruit group
Other: Nipple group — Nipple Stimulation
  Arms: Nipple group

SUMMARY:
The study was conducted to determine the effect of consumption of date fruit and nipple stimulation on labor.

The samples were applied to pregnant women satisfying the research criteria in a state hospital in Istanbul between October 2013 and June 2014.

DETAILED DESCRIPTION:
The study was designed to be randomly controlled. Block randomization method was used to determine the experimental and control groups. Randomization was done by a biostatistician outside the researcher. 198 pregnant women were randomly assigned to the date fruit, nipple and control groups. From the 37th gestational age to the onset of labor, 6 date fruits were consumed per day by the date fruit group and the nipple stimulation was applied 6 minutes per day for the nipple group. No intervention was made for the control group. For the collection of research data, "Structured Information Form" and "Wijma Birth Expectancy / Experience Scale Version" were used.

ELIGIBILITY:
Inclusion Criteria:

* Women who nulliparous at the 37th gestational age, have singleton pregnancy, have the BMI is less than 25 kg/m2, planning to have a normal vaginal delivery, have vertex presentation, a volunteer to participate in the study, no smoking in pregnancy and have moderate birth fear according to W-DEQ were included in the study.

Exclusion Criteria:

* Women who have risk pregnancy (such as preterm labor risk, preeclampsia eclampsia, premature rupture of membranes, placenta previa, gestational diabetes, fetal anomaly and chronic diseases) were excluded in the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant Women
Enrollment: 198 (Actual)
Dates: Start 2013-10-10 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
The spontaneous onset of labor | From the 37th gestational age to the labor
  The spontaneous onset of labor (dichotomous data: yes or no)
Induction and augmentation of labor | From the 37th gestational age to the labor
  Induction and augmentation of labor (dichotomous data: yes or no)

SECONDARY OUTCOMES:
Mode of delivery | From the 37th gestational age to the birth
  Mode of delivery (dichotomous data: vaginal delivery or caesarean section)

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Rathfisch, Prof, Study Director — Atlas University
Locations (1):
- Zeynep Kamil Women's and Children's Diseases Training and Research Hospital, Istanbul, Turkey (Türkiye)